CLINICAL TRIAL: NCT05507242
Title: Effects of Blocking TSLP on Airway Inflammation and the Epithelial Immune-response to Exacerbation Triggers in Patients With COPD A Randomized Double-blind, Placebo-controlled Trial of Tezepelumab UPSTREAM-COPD
Brief Title: Effects of Blocking TSLP on Airway Inflammation and the Epithelial Immune-response to Exacerbation Triggers in Patients With COPD
Acronym: UPSTREAM-COPD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Asger Sverrild (Other)
Collaborators: AstraZeneca (Industry); University Hospitals, Leicester (Other)
Responsible Party: Sponsor-Investigator, Asger Sverrild, MD, PhD, Clinical Associate Professor, Bispebjerg Hospital
Organization: Bispebjerg Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UPSTREAM-COPD
Record Dates: First submitted 2022-08-17; First posted 2022-08-18 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: COPD; COPD Exacerbation; COPD Bronchitis; Airway Disease; Immune System Disorder
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Immune System Diseases | interventions — tezepelumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tezepelumab (Experimental): Tezepelumab subcutaneous injection
  Interventions: Biological: Tezepelumab
- Placebo (Placebo Comparator): Placebo subcutaneous injection
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Tezepelumab — Tezepelumab 210 mg for 20 weeks (5 doses in total, 4-week intervals), administered subcutaneously
  Arms: Tezepelumab
Other: Placebo — Placebo subcutaneous injection for 20 weeks (5 doses in total, 4-week intervals)
  Arms: Placebo

SUMMARY:
A phase 2, multicentre, randomized, double-blind, placebo-controlled, parallel group study to evaluate the effect of tezepelumab on airway inflammation in patients with COPD.

DETAILED DESCRIPTION:
This is a multicentre, randomized, double-blind, placebo-controlled, parallel group study to evaluate the effect of tezepelumab on airway inflammation in patients with COPD on LABA+LAMA±ICS with ≥ 1 exacerbation the past 12 months. Approximately 80 subjects will be randomized to receive tezepelumab, or placebo, administered via subcutaneous injection at the study site, over a 20-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* A diagnosis of COPD (according to GOLD (GOLD 2021 Report))
* ≥ 10 packyears smoked (current or ex-smokers)
* Age 40 years or older
* Postbronchodilator FEV1 ≥ 30% predicted (and ≥ 1.0L) and < 80% predicted
* Maintenance treatment with LAMA+LABA±ICS (stable dose) for at least 3 months prior to V1
* ≥1 prednisolon and/or antibiotic treated exacerbation in the past 12 months
* Subjects must demonstrate acceptable inhaler and spirometry techniques during screening (as evaluated and in the opinion of study site staff)
* Subjects must demonstrate ≥ 70% compliance with daily inhalers during the screening/run-in
* Females of childbearing potential who are sexually active with a nonsterilized male partner must use a highly effective method of contraception from the time informed consent is obtained and must agree to continue using such precautions through Week 20 of the study; cessation of contraception after this point should be discussed with a responsible physician. Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception. Females of childbearing potential are defined as those who are not surgically sterile (ie, bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or postmenopausal (defined as 12 months with no menses without an alternative medical cause).

Exclusion Criteria:

* Previous medical history or evidence of an uncontrolled intercurrent illness that in the opinion of the investigator may compromise the safety of the subject in the study or interfere with evaluation of the investigational product or reduce the subject's ability to participate in the study. Subjects with well-controlled comorbid disease (eg, hypertension, hyperlipidemia, gastroesophageal reflux disease) on a stable treatment regimen for 15 days prior to Visit 1 are eligible.
* Any concomitant respiratory disease that in the opinion of the investigator will interfere with the evaluation of the investigational product or interpretation of subject safety or study results (e.g., cystic fibrosis, pulmonary fibrosis, aspergillosis, active tuberculosis).
* Current asthma
* Lung volume reduction surgery for COPD
* Exacerbation requiring oral corticosteroids or antibiotics (any dose for more than 3 days) 4 weeks prior to Visit 1 or during the run-in period
* Any use of home oxygen therapy
* Any clinically relevant abnormal findings in hematology or clinical chemistry (laboratory results from Visit 1), physical examination, vital signs during the screening, which in the opinion of the investigator, may put the subject at risk because of his/her participation in the study, or may influence the results of the study, or the subject's ability to participate in the study
* History of cancer: Subjects who have had basal cell carcinoma or in situ carcinoma of the cervix are eligible to participate in the study provided that curative therapy was completed at least 12 months prior to Visit 1. Subjects who have had other malignancies are eligible provided that curative therapy was completed at least 5 years prior to Visit 1.
* Acute upper or lower respiratory infections requiring antibiotics or antiviral medications within 4 weeks prior to Visit 1 or during the screening period
* A positive human immunodeficiency virus (HIV) test at screening or subject taking antiretroviral medications, as determined by medical history
* Positive hepatitis B surface antigen, or hepatitis C virus antibody serology at screening, or a positive medical history for hepatitis B or C. Subjects with a history of hepatitis B vaccination without history of hepatitis B are allowed to enroll.
* History of sensitivity to any component of the investigational product formulation or a history of drug or other allergy that, in the opinion of the investigator or medical monitor contraindicates their participation.
* History of any known primary immunodeficiency disorder excluding asymptomatic selective immunoglobulin A or IgG subclass deficiency.
* Active tuberculosis or history of untreated latent tuberculosis
* History of anaphylaxis to any biologic therapy.
* Use of immunosuppressive medication (eg, methotrexate, troleandomycin, oral gold, cyclosporine, azathioprine, intramuscular long-acting depot corticosteroid, or any experimental anti-inflammatory therapy) within 3 months prior to Visit 1.
* Receipt of any of the following within 30 days prior to Visit 1: immunoglobulin or blood products, or receipt of any investigational nonbiologic agent within 30 days or 5 half-lives prior Visit 1, whichever is longer.
* Receipt of any marketed or investigational biologic agent within 4 months or 5 half- lives prior to Visit 1, whichever is longer.
* Pregnant, breastfeeding or lactating females
* History of chronic alcohol or drug abuse within 12 months prior to Visit 1.
* Planned surgical procedures requiring general anesthesia or in-patient status for > 1 day during the conduct of the study.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Concurrent enrollment in another clinical study involving an investigational treatment.
* Receipt of any live or attenuated vaccines within 15 days prior to Visit 1.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-10-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect of tezepelumab on eosinophilic bronchial mucosal tissue inflammation | 20 weeks
  The change, expressed as ratio, in eosinophil cell counts per mm2 from baseline to week-20

SECONDARY OUTCOMES:
To evaluate the effect of tezepelumab on neutrophilic bronchial mucosal tissue inflammation | 20 weeks
  The change, expressed as ratio, in neutrophil cell couts per mm2 from baseline to week-20
To evaluate the effect of tezepelumab on mast cell bronchial mucosal tissue inflammation | 20 weeks
  The change, expressed as ratio, in mast cell couts per mm2 from baseline to week-20
To evaluate the effect of tezepelumab on CD4+ cell bronchial mucosal tissue inflammation | 20 weeks
  The change, expressed as ratio, in CD4+ cell couts per mm2 from baseline to week-20
To evaluate the effect of tezepelumab on CD8+ cell bronchial mucosal tissue inflammation | 20 weeks
  The change, expressed as ratio, in CD8+ cell couts per mm2 from baseline to week-20
To evaluate the effect of tezepelumab on macrophage cell bronchial mucosal tissue inflammation | 20 weeks
  The change, expressed as ratio, in macrophage cell couts per mm2 from baseline to week-20

CONTACTS AND LOCATIONS:
Overall Officials: Asger Sverrild, MD, PhD, Principal Investigator — Bispebjerg Hospital
Locations (2):
- Research site, Copenhagen, Denmark
- Research site, Leicester, United Kingdom